CLINICAL TRIAL: NCT02543606
Title: A Randomized, Two-way Crossover, Single-dose Pharmacokinetic Study to Evaluate the Bioequivalence of Esomelone for Injection/Infusion (Esomeprazole 40mg), Compared to Reference Drug (Nexium 40mg) in Healthy Adult Subjects
Brief Title: Bioequivalence of Two Formulations of Esomeprazole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Collaborators: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YSP-RFH3002-01
Record Dates: First submitted 2015-08-24; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esomelone (Experimental): powder for injection/ infusion Esomeprazole 40mg
  Interventions: Drug: Esomelone; Drug: Nexium
- Nexium (Active Comparator): powder for injection/ infusion Esomeprazole 40mg
  Interventions: Drug: Esomelone; Drug: Nexium

INTERVENTIONS:
Drug: Esomelone — powder for injection/ infusion Esomeprazole 40mg
Drug: Nexium — powder for injection/ infusion Esomeprazole 40mg

SUMMARY:
Bioequivalence of Two Formulations of Esomeprazole 40mg

DETAILED DESCRIPTION:
A randomized, two-way crossover, single-dose pharmacokinetic study to evaluate the bioequivalence of a test formulation of Esomelone powder for solution for injection/infusion 40mg (Esomeprazole 40mg), compared to an equivalent dose of a reference drug product (Nexium powder for injection and infusion 40mg) in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult, aged between 20 to 40 years old.
2. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, laboratory tests, chest x-ray and electrocardiogram.

   * no particular clinical significance in clinical examination and laboratory tests within two months (60 days) prior to Period I dosing.
   * normal or considered not clinically significant by the investigator chest X-ray and ECG results within six months (180 days ) prior to Period I dosing.
3. The normal range of the body mass index should be between 18.5 and 25; body mass index equals [weight (kg)]/[height (m)]2.
4. Normal laboratory determinations result (within normal range or considered not clinically significant by the investigator) including: SGOT (AST), SGPT (ALT), albumin, glucose, creatinine, uric acid, cholesterol, TG, r-GT, alkaline phosphatase, total bilirubin, BUN, HBsAg, Anti-HCV and Anti-HIV test.
5. Normal hematology results (within normal range or considered not clinically significant by the investigator) including: hemoglobin, hematocrit, WBC count with differential, RBC count and platelet count.
6. Normal urinalysis results (within normal range or considered not clinically significant by the investigator) including: glucose, protein, RBC, WBC, epith, casts and bacteria.
7. Female subject who is

   * using adequate contraception since last menstruation and no plan for conception during the study,
   * non-lactating.
   * has negative pregnancy test (urine) within 14 days prior to the study.
8. Informed consent form signed.

Exclusion Criteria:

1. A history of drug or alcohol abuse during the past 24 weeks.
2. Sensitivity to analogous drug.
3. A clinically significant illness (such as significant unintentional weight loss, recurrent vomiting, dysphagia, haematemesis, melaena or gastric ulcer) within the past 4 weeks.
4. Evidence of any clinical significant renal, cardiovascular, hepatic, hematopoietic, neurological, pulmonary or gastrointestinal pathology within the past 4 weeks.
5. Planned vaccination during the time course of the study.
6. Participation of ant clinical investigation during the last 60 days.
7. Regular use of any medication during the last 4 weeks.
8. Single use of any medication during the last 2 weeks.
9. Blood donation of more than 250 mL within the past 12 weeks.
10. Individuals are judged by the investigation or co-investigator to be undesirable as subjects.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic parameters of ln transformed data ln(AUC) of the product. | pre-dose to 12 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Zen Yeh, M.D., Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan